CLINICAL TRIAL: NCT03121196
Title: Social Deprivation and Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-319; 2016-A02076-45 (Other: 2016-A02076-45)
Record Dates: First submitted 2017-04-14; First posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Gestational Diabetes; High Blood Pressure; Prematurity; Fetal Growth Restriction
Keywords: Social deprivation; Adverse perinatal outcomes
MeSH Terms: conditions — Diabetes, Gestational; Hypertension; Premature Birth; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- deprived women: Two groups of women will be compared deprived women and non-deprived women
  Interventions: Other: Epices score
- non-deprived women: Two groups of women will be compared deprived women and non-deprived women
  Interventions: Other: Epices score

INTERVENTIONS:
Other: Epices score — Association between EPICES score and the adverse perinatal outcomes will be assessed by quantile regression

SUMMARY:
Social deprivation during pregnancy is associated to adverse perinatal outcomes. However, prenatal screening of social deprivation by reliable measurement is not performed. Prevalence of social deprivation is yet underestimated during pregnancy and vulnerable women are not being provided optimal prenatal care.

Our aim is to validate EPICES score during pregnancy.

DETAILED DESCRIPTION:
The process of deprivation was defined first by J. Wrezinski and P. Townsend who also reported that deprivation is the main cause of inequalities in health. Several studies have already shown an association between socioeconomic deprivation and adverse birth outcomes. EPICES score is the only one that measure individual deprivation. The EPICES score should be therefore included systematically in standard follow-up of pregnant women.

Descriptive analysis will assess women's characteristics and prevalence of social deprivation. Two groups of women will be compared deprived women and non-deprived women.

Association between EPICES score and the adverse perinatal outcomes will be assessed by quantile regression.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* delivery at 2 maternity hospitals of Clermont-Ferrand area
* fluent command of spoken and written French

Exclusion Criteria:

* Terminations of pregnancy
* protected women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 615 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Epices score distribution | at day 1
  Association between EPICES score and the adverse perinatal outcomes will be assessed by quantile regression

SECONDARY OUTCOMES:
Adverse perinatal outcomes | at day 1
  Association between EPICES score and the adverse perinatal outcomes will be assessed by quantile regression

CONTACTS AND LOCATIONS:
Overall Officials: Françoise VENDITELLI, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France